CLINICAL TRIAL: NCT00076596
Title: Brain Reorganization in Cerebral Palsy
Brief Title: Brain Control of Movements in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040098; 04-N-0098
Record Dates: First submitted 2004-01-26; First posted 2004-01-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Cerebral Palsy
Keywords: Corticospinal Tracts; Spastic Hemiplegia; Spastic Diplegia; Cortical Re-Organization; Functional Outcome; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

SUMMARY:
This study will examine how the brain controls movements in patients with certain types of cerebral palsy. In healthy people, one side of the body usually controls movements on the other side of the body. In patients with cerebral palsy, this pattern may be altered, and one side of the brain may control movements on the same side of the body. Information obtained from this study may lead to improved rehabilitation therapy strategies for patients with cerebral palsy.

Healthy volunteers and patients with cerebral palsy between 6 and 18 years of age may be eligible for this study. All candidates will be screened with a medical history, physical examination, and psychological testing. In addition, patients with cerebral palsy will have hearing and vision tests, a review of their medical records, and a magnetic resonance imaging (MRI) scan if one has not been done within the past year. For this test, the patient lies on a table that slides into a narrow metal cylinder with a strong magnetic field (the scanner). The scanning time usually lasts between 45 and 90 minutes.

Patients enrolled in the study also will be evaluated by a physiatrist and physical and occupational therapists. They will be examined for muscle stiffness and reflexes. Their gait and movements (e.g., how they pick up a glass of water) will be evaluated. They will be asked about their ability to perform activities around the house and at school and whether a wheelchair or walker is needed to get around. Patients may also be asked about how they are dealing with their movement problems and how it affects their caregivers.

All participants will undergo three tests, described below, to evaluate movement control. The first two tests use electrodes (small metal discs) taped to the skin over the muscles in both hands to measure muscle activity. A small disc placed on the fingers detects and measures the hand movements. The third test uses magnetic pulses that stimulate the brain to study how the brain controls movements.

1. Quantitative test of fine motor function: For this test, the subject taps buttons at different speeds on a box attached to a computer. The test is similar to playing simple computer games.
2. Long latency reflexes: For this test, the subject's hand is lightly strapped into a holder that holds the hand still while a motor moves the index finger with sudden small movements. These reflexes may also be tested using a gentle shock to the finger delivered through a ring electrode.
3. Transcranial magnetic stimulation: For this test, the subject sits in a comfortable chair. An insulated coil is held on the scalp. A magnetic pulse from the coil stimulates the brain. The subject may hear a click and feel a snap or pulling sensation on the scalp under the coil. The stimulation may also cause twitching in the muscles of the arm or leg. During the stimulation, the subject may be asked to move certain muscles or perform other simple actions.

DETAILED DESCRIPTION:
Although the capacity of the immature nervous system to recover after injury is superior to that of the adult brain, children with cerebral palsy carry a great burden of morbidity for their entire life. Functional outcome may be determined not only by characteristics of the lesion (size, location, and timing) but also by the response of the brain to the lesion (cortical re-organization). Little is known about how underlying limitations, such as inefficient cortical re-organization, affect functional outcome and response to therapy in children with cerebral palsy. Because of this, individual rehabilitation strategies are based solely on the level of functioning rather than on the underlying impairment. Research demonstrates that novel rehabilitation strategies can manipulate plasticity of the motor cortex and, in this way, improve functional outcome in adults who have suffered a stroke. There is preliminary evidence that these treatments may also benefit patients with cerebral palsy. However, cortical re-organization after an injury to the developing brain may not be similar to that which occurs after a stroke in the adult brain. It would be of benefit to have a greater understanding of the impairments that arise from inefficient cortical re-organization in children with cerebral palsy. It is also important to have the research methodology to assess the effect of these novel treatments in order to measure their true benefit.

Cortical re-organization can lead to enhanced participation of the unaffected hemisphere via anomalous ipsilateral corticofugal motor projections. Recent evidence suggests that this form of neural re-organization may not be efficient. Three different types of ipsilateral projections are thought to exist: 1) fast-conducting developmental ipsilateral projections that persist beyond the age at which they normally disappear; 2) slow-conducting ipsilateral tracts present in healthy subjects that become more accessible after injury; 3) fast-conducting projections that arise de novo from the ipsilateral primary motor cortex after injury to the developing brain. Each type has a distinct neurophysiologic profile that can be characterized using transcranial magnetic stimulation (TMS) and electromyography (EMG).

To date, the relationship between anomalous ipsilateral corticofugal motor projections and functional outcome has not been examined in detail. There is preliminary evidence that the presence of these anomalous ipsilateral projections is associated with poor outcome, suggesting that they represent an inefficient cortical re-organization process. In addition, the anomalous projections that arise de novo from the ipsilateral primary motor cortex appear to have the worst prognosis. The proposed research study will characterize anomalous ipsilateral corticofugal motor projections in a group of children with spastic hemiplegia and spastic diplegia subtypes of cerebral palsy using TMS and EMG. We will evaluate functional limitations of the hand in these children and will examine the relationship between each type of ipsilateral pathway and functional outcome. In this way, it will be possible to determine which anomalous ipsilateral projections are associated with poor function in patients with cerebral palsy.

This study will increase our understanding of the functional significance of these ipsilateral projections and will make it possible to identify these ipsilateral projections in individual children. The neurophysiologic techniques developed in this study will provide essential research methodology to assess brain re-organization before and after novel therapeutic approaches.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children and adults 6 to 30 years of age.

CEREBRAL PALSY PATIENTS:

Patients previously diagnosed with spastic diplegia or spastic hemiplegia subtype of cerebral palsy.

Lesions must be pre-, peri- or post-natal and acquired before 1 year of age.

Lesions must be non-progressive.

Patients must be able to voluntarily move their upper and lower limbs.

Cognitive function: DQ over 50 or IQ over 50 as assessed by Gesell or with standardized tests (pre-school age), or through school testing (school age).

Able to attend, at minimum, one-on-one tutoring or special education classes (to ensure cooperation with testing procedures).

Able to ambulate either independently or with assistive mobility devices.

HEALTHY SUBJECTS:

Scores below 60 on Connor's (ADHD) checklist.

Normal neurological history and examination.

EXCLUSION CRITERIA:

Any child who is pregnant. Adult women and girls between 12 and 17 years of age who have started their menstrual periods will be required to take a pregnancy test at the initial interview. If this is positive, they will not be allowed to take part in the study. At the initial phone screening we will inform both the parent/ guardian and the child that we will require this pregnancy test at the initial interview to determine eligibility and that we will inform both the child and her parents with the results of the test.

CEREBRAL PALSY PATIENTS:

Patients with subtypes of cerebral palsy that are not hemiplegia or diplegia. These include spastic quadriplegia (no difference in level of severity of motor deficit between arms and legs); spastic triplegia; mixed forms of cerebral palsy; athetoid or dystonic forms of cerebral palsy; unclassifiable forms of cerebral palsy.

Hemiplegic cerebral palsy with greater than minimal motor deficits on the good hand.

Spastic diplegia patients who have asymmetry of the motor deficit greater than 1 severity point between the two sides (e.g. left side mild, right side severe).

Patients with DQ or IQ below 50 as assessed by Gesell or with standardized tests (pre-school age), or through school testing (school age).

Uneducable patients by reason of severely impaired attention.

Patients with seizures within the last 6 months.

Patients with an underlying known genetic or chromosomal disorder.

Patients with clearly identified familial or non-familial syndromes (without known chromosomal or genetic defect).

Cerebral lesions acquired after 1 year of age.

Patients with progressive or neurodegenerative disorders.

Patient with spinal disorders in the absence of cerebral lesions.

Patients with cerebral lesions caused by sickle cell disease or by emboli associated with congenital cardiac lesions.

Patients with severe cognitive deficits who cannot follow simple verbal commands.

Patients incapable of voluntary movement of either upper or lower limbs due to contractures.

Patients who have had rhizotomy for upper extremity plasticity, who have had botulinum toxin within the last 3 months or have an intrathecal baclofen pump.

Patients with severe postural abnormalities who cannot maintain supported sitting.

HEALTHY SUBJECTS:

Children or adults with any neurological and/or psychiatric disorder including attention deficit hyperactivity disorder or learning disorder.

Subjects with any chronic medical disorders.

Subjects taking regular medications, including medications for allergies, hormonal oral contraceptives, or over-the-counter medications.

Healthy subjects born before 36 weeks gestation as estimated by dates, ultrasound or other methods (if a discrepancy exists, then the ultrasound estimation will be taken as definitive).

Subjects with siblings who have developmental delay or abnormalities of the corpus callosum (these subjects have an increased chance of having asymptomatic abnormalities of the central nervous system).

Subjects with albinism or a personal or family history of sensorineural hearing loss (these subjects have an increased incidence of incidental callosal abnormalities).

EXCLUSIONARY CRITERIA FOR CLINICAL MRI STUDIES:

Any subject with metal objects in the body such as pacemakers, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses, cochlear implants, or shrapnel fragments).

Any subject with permanent tattoos on the eyelids (ferromagnetic (iron oxide-based) tattoo pigments can interact with the static magnetic field of an MRI imager).

Any subject that would require sedation for the scan.

EXCLUSIONARY CRITERIA FOR TMS:

Cerebral palsy patients on neuroactive medications (e.g. antiepileptics).

Patients with hearing loss (greater than 15 dB at any individual frequency) in either ear (as evaluated in the Audiology Department, CC, NIH).

Healthy children with a personal history of febrile seizures and with a family history of first degree relatives with seizures.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130
Dates: Start 2004-01-23; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Georgetown University Medical Center, Washington D.C., District of Columbia

REFERENCES:
- [Background] Staudt M, Grodd W, Gerloff C, Erb M, Stitz J, Krageloh-Mann I. Two types of ipsilateral reorganization in congenital hemiparesis: a TMS and fMRI study. Brain. 2002 Oct;125(Pt 10):2222-37. doi: 10.1093/brain/awf227. PMID 12244080